CLINICAL TRIAL: NCT04000529
Title: A Phase Ib, Open-label, Multi-center Study to Characterize the Safety, Tolerability, and Preliminary Efficacy of TNO155 in Combination With Spartalizumab or Ribociclib in Selected Malignancies
Brief Title: Phase Ib Study of TNO155 in Combination With Spartalizumab or Ribociclib in Selected Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTNO155B12101
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Carcinoma; Head and Neck Squamous Cell Carcinoma; Esophageal SCC; Gastrointestinal Stromal Tumors; Colorectal Cancer
Keywords: TNO155, spartalizumab, ribociclib, checkpoint inhibitor, SHP2, PD-1, CDK4/6, NSCLC, CRC, HNSCC, KRAS, esophageal SCC, GIST
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma; Gastrointestinal Stromal Tumors; Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — spartalizumab; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNO155 in combination with spartalizumab (Experimental): TNO155 in combination with spartalizumab
  Interventions: Drug: TNO155; Drug: Spartalizumab
- TNO155 in combination with ribociclib (Experimental): TNO155 in combination with ribociclib
  Interventions: Drug: TNO155; Drug: Ribociclib

INTERVENTIONS:
Drug: TNO155 — Capsule
Drug: Spartalizumab — Concentrate for solution for infusion
  Other Names: PDR001
  Arms: TNO155 in combination with spartalizumab
Drug: Ribociclib — Capsule and tablet
  Other Names: LEE011
  Arms: TNO155 in combination with ribociclib

SUMMARY:
This study was a Phase Ib, multi-center, open-label study of TNO155 in combination with spartalizumab or ribociclib with a dose escalation part followed by a dose expansion part in adult subjects with advanced solid tumors.

These two treatment arms enrolled subjects in parallel to characterize the safety, tolerability, PK, PD and preliminary antitumor activity.

The study treatment was administered until the subject experienced unacceptable toxicity, progressive disease, and/or had treatment discontinued at the discretion of the Investigator or the subject, or due to withdrawal of consent.

DETAILED DESCRIPTION:
Rationale The purpose of this study was to evaluate the safety, tolerability, and preliminary efficacy of the combination of TNO155 with spartalizumab and of TNO155 with ribociclib, and to identify dosing regimens for further study. Data from preclinical models have demonstrated anti-tumor activity for the combinations of TNO155 with spartalizumab and of TNO155 with ribociclib that is superior to the activity observed with each of the drugs as single agents. These data suggest that these combinations may provide clinical benefit to patients with advanced malignancies.

Study Design This study was a Phase Ib, multi-center, open-label study with a dose escalation part followed by a dose expansion part in adult subjects with advanced solid tumors to characterize the safety and tolerability TNO155 in combination with spartalizumab and of TNO155 in combination with ribociclib and to identify the MTD and/or recommended regimen (dose and schedule) for each combination. The study treatment was administered until the subject experienced unacceptable toxicity, progressive disease, and/or had treatment discontinued at the discretion of the Investigator or the subject, or due to withdrawal of consent.

Objectives

Primary objective:

To characterize the safety and tolerability TNO155 in combination with spartalizumab and of TNO155 in combination with ribociclib, and to identify the MTD and/or recommended regimen (dose and schedule) for each combination.

Secondary objectives:

* To characterize the pharmacokinetic (PK) profile of TNO155, spartalizumab and ribociclib when administered as a combination of TNO155 plus spartalizumab or of TNO155 plus ribociclib.
* To evaluate the preliminary anti-tumor activity of TNO155 in combination with spartalizumab and of TNO155 in combination with ribociclib.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Age ≥ 18 years. For Japan only: written consent is necessary both from the patient and his/her legal representative if he/she is under the age of 20 years.
3. ECOG (Eastern Cooperative Oncology Group) performance status ≤ 1.
4. Dose escalation part: Patients with advanced solid tumors, with evaluable disease as determined by RECIST version 1.1, and fit into one of the following groups:

   a. For TNO155 plus spartalizumab combination: i. Advanced EGFR WT, ALK WT NSCLC, after progression on or intolerance to platinum-containing combination chemotherapy and after progression on anti-PD-1 or anti-PD-L1 therapy.

   ii. Advanced HNSCC or esophageal SCC, after progression on or intolerance to platinum-containing combination chemotherapy.

   iii. Advanced CRC, after progression on or intolerance to all standard-of-care (SOC) therapy per local guidelines.

   b. For TNO155 plus ribociclib combination: Advanced solid malignancies with the exception of CRC or GIST, after progression on or intolerance to all SOC therapy per local guidelines. The exclusion of CRC applies only as of Protocol Amendment 4.
5. Dose expansion part: Patients with advanced solid tumors, with at least one measurable lesion as determined by RECIST version 1.1, who fit into one of the following groups:

   a. For TNO155 plus spartalizumab combination: i. Advanced EGFR WT, ALK WT, KRAS G12C NSCLC after progression on or intolerance to platinum-containing combination chemotherapy and after progression on anti-PD-1 or anti-PD-L1 therapy.

   ii. Advanced EGFR WT, ALK WT, KRAS WT NSCLC, after progression on or intolerance to platinum-containing combination chemotherapy and after progression on anti-PD-1 or anti-PD-L1 therapy.

   iii. Advanced HNSCC, after progression on or intolerance to, platinum-containing combination chemotherapy.

   b. For TNO155 plus ribociclib combination: i. Advanced EGFR WT, ALK WT, KRAS WT NSCLC, after progression on or intolerance to platinum-containing chemotherapy and anti-PD-1 or anti-PD-L1 therapy ii. Advanced HNSCC, after progression on or intolerance to all SOC per local guidelines
6. Patients with NSCLC whose tumors harbor genomic aberrations for which SOC targeted therapies exist and are locally approved and available must have had progression on or after, or intolerance to, the SOC targeted therapy/therapies as indicated
7. Patients must have a site of disease amenable to biopsy

Key Exclusion Criteria:

1. Prior treatment with a MAPK pathway inhibitor
2. Clinically significant cardiac disease or risk factors
3. Use of any agent known to prolong the QT interval unless it can be permanently discontinued for the duration of study (see list in Section 6.2.2).
4. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO
5. Inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drugs
6. Symptomatic CNS metastases which are neurologically unstable
7. Insufficient bone marrow function at screening:

   1. Absolute Neutrophil Count (ANC) < 1.5 x 109/L.
   2. Hemoglobin < 9.0 g/dL.
   3. Platelets < 75 x 109/L for TNO155 plus spartalizumab combination; < 100 x 109/L for TNO155 plus ribociclib combination.
8. Insufficient hepatic or renal function at screening:

   1. Serum total bilirubin > upper limit of normal (ULN) or, for TNO155 plus spartalizumab combination only, if liver metastases are present at baseline, serum total bilirubin > 1.5 x ULN. An exception for either combination is for patients with Gilbert's syndrome, who are excluded if total bilirubin > 3.0 x ULN or direct bilirubin > 1.5 x ULN
   2. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x ULN for TNO155 plus spartalizumab combination or > 2.5 x ULN for TNO155 plus ribociclib combination, or > 5 x ULN for either combination if liver metastases are present.
   3. Creatinine clearance < 60 mL/min (calculated using Cockcroft-Gault equation).
9. Pregnant or breast-feeding (lactating) women.

   Additional exclusion criteria for the TNO155 plus spartalizumab combination
10. History of severe hypersensitivity reactions to other mAbs.
11. Active, known or suspected autoimmune disease.
12. History of or current interstitial lung disease or pneumonitis grade ≥ 2.
13. Human Immunodeficiency Virus (HIV) infection, unless the patient is on antiviral therapy and has undetectable viral load.
14. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
15. Systemic chronic steroid therapy
16. Patients who discontinued prior anti-PD-1 therapy due to an anti-PD-1-related toxicity.

    Additional exclusion criteria for the TNO155 plus ribociclib combination
17. Systolic Blood Pressure (SBP) < 90 mmHg.
18. International Normalized Ratio (INR) > 1.5 (unless the patient is receiving anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within seven days prior to the first dose of study drug).
19. History of HIV infection (testing not mandatory)
20. Currently receiving any of the following substances and cannot be discontinued seven days prior to Cycle 1 Day 1:

    * Concomitant medications or herbal supplements, that are strong inducers or inhibitors of CYP3A4/5,
    * Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
21. Previous treatment with a CDK4/6 inhibitor.
22. Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment.

Note: The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
DLT incidence | 1 year
  Incidence of dose limiting toxicities (DLTs) during the first cycle of combination treatment during the dose escalation part
AE and SAE incidence | 3 years
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as per CTCAE v5.0, by treatment
Dose interruptions, reductions and dose intensity, by treatment | 3 years
  Dose tolerability

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Cmax | 3 years
  Cmax for TNO155, spartalizumab, and ribociclib
Pharmacokinetics (PK): Tmax | 3 years
  Tmax for TNO155, spartalizumab, and ribociclib
Pharmacokinetics (PK): AUClast | 3 years
  AUClast for TNO155, spartalizumab, and ribociclib
Pharmacokinetics (PK): AUCtau | 3 years
  AUCtau for TNO155, spartalizumab, and ribociclib
Efficacy measurements per RECIST v1.1: ORR | 3 years
  Overall response rate (ORR) per RECIST v1.1, by treatment
Efficacy measurements per RECIST v1.1: DCR | 3 years
  Disease control rate (DCR) per RECIST v1.1, by treatment
Efficacy measurements per RECIST v1.1: PFS | 3 years
  Progression-free survival (PFS) per RECIST v1.1, by treatment
Efficacy measurements per RECIST v1.1: DOR | 3 years
  Duration of response (DOR) per RECIST v1.1, by treatment
Efficacy measurements per iRECIST: ORR | 3 years
  Overall response rate (ORR) per iRECIST for TNO155 in combination with spartalizumab
Efficacy measurements per iRECIST: DCR | 3 years
  Disease control rate (DCR) per iRECIST for TNO155 in combination with spartalizumab
Efficacy measurements per iRECIST: PFS | 3 years
  Progression-free survival (PFS) per iRECIST for TNO155 in combination with spartalizumab
Efficacy measurements per iRECIST: DOR | 3 years
  Duration of response (DOR) per iRECIST for TNO155 in combination with spartalizumab
Overall Survival | 3 years
  Overall survival (OS) by treatment

CONTACTS AND LOCATIONS:
Locations (10):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Novartis Investigative Site, Westmead, New South Wales, Australia
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Chengdu, Sichuan, China
- Novartis Investigative Site, Cologne, Germany
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen H, Cresswell GM, Libring S, Ayers MG, Miao J, Zhang ZY, Solorio L, Ratliff TL, Wendt MK. Tumor Cell-Autonomous SHP2 Contributes to Immune Suppression in Metastatic Breast Cancer. Cancer Res Commun. 2022 Oct 3;2(10):1104-1118. doi: 10.1158/2767-9764.CRC-22-0117. eCollection 2022 Oct. PMID 36969745
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18246
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2476